CLINICAL TRIAL: NCT05411003
Title: Is Nottingham Extended Activities Of Daily Living Scale in Urdu Language a Reliable and Valid Tool to Assess the Level of Independence While Performing Activities of Daily Livings
Brief Title: Urdu Version Of Nottingham Extended Activities Of Daily Living Scale: Reliability And Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00270
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Nottingham Extended Activities Of Daily Living Scale; Urdu Version; Reliability; Validity; Stroke; Neurological Disorders; Activities of Daily Living
MeSH Terms: conditions — Stroke; Nervous System Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to know the validity and reliability as well as to translate and culturally adapt the Nottingham Extended Activities Of Daily Living Scale into Urdu language in Pakistani population of Stroke. This study also aims to correlate the scale with the Modified Barthel Index and Frenchay Activities Index.

DETAILED DESCRIPTION:
As per previous recommendation the English version of Nottingham Extended Activities Of Daily Living Scale will be translated into Urdu and it will be culturally adapted. Nottingham Extended Activities Of Daily Living Scale will be given to eighty individuals of stroke population which were selected on the basis of convenience sampling and the criteria of inclusion and exclusion. Study will investigate both inter-observer and intra-observer reliability of Nottingham Extended Activities Of Daily Living Scale, Modified Barthel Index and Frenchay Activities Index; the 2 set of questionnaire designed will be given to the participants on the same day to be filled, by two observers. And with a gap of half an hour between distributions of first two forms questionnaires will be given for inter-observer assessment. And after a time period of one week a third assessment will be collected by the first observer (intra-observer assessment). Statistical Package of Social Sciences Version 24 will be used for data entry and analysis. Cronbach alpha value will be used for checking internal consistency and intra-class correlation coefficient will be used to analyze test retest reliability.

ELIGIBILITY:
Inclusion Criteria:

1. Having age of 67 years or more
2. Having stroke
3. Both males and females

Exclusion Criteria:

1. Neurological condition other than stroke
2. Any fracture of lower extremity
3. Any amputation of lower extremity

Min Age: 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Stroke population of Pakistan over 67 years of age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Nottingham Extended Activities Of Daily Living Scale | 1st day
  The purpose of development of Nottingham Extended Activities Of Daily Living Scale was to use it for stroke patients. Each question on the scale is graded either 0 which means patient cannot perform task, 1 which means that patient can do activity but with assistance, 2 which states that task can be performed but with difficulty, 3 which means that he or she can perform the activity on his or her own easily. The score ranges from 0-66.
Frenchay Activities Index | 1st day
  The Frenchay Activities Index is a tool for assessing instrumental activities of daily living in stroke patients. It is based upon the frequency in which activities are performed. Frenchay Activities Index scores vary from 0 (inactive) to 45 (very active), with 0-15 indicating inactivity, 16-30 indicating moderate activity, and 31-45 indicating extreme activity. A score of 18 or more than 18 was used to predict minor impairment following a stroke.
Modified Barthel Index | 1st day
  The Barthel modified index scale is used to assess behavior related to daily tasks in stroke patients or those with other debilitating conditions. Each activity is given a score ranging from 0 (unable to complete task) to 5, 10, or 15 (highest) (fully independent- exact score depends on the activity being evaluated). Summing the scores for each of the items yields a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No